CLINICAL TRIAL: NCT07219888
Title: Comparison of Suzetrigine and Oxycodone for Postoperative Pain and Analgesic Requirements After Primary Total Knee Arthroplasty: a Prospective, Randomized Study
Brief Title: Comparison of Suzetrigine and Oxycodone for Postoperative Pain After Primary Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Clinical Professor, Chief, Adult Reconstruction, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25.0688
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; knee; total knee arthroplasty; prospective RCT; postoperative analgesia; postoperative pain management
MeSH Terms: conditions — Osteoarthritis | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Prospective, randomized cohort analysis study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: suzetrigine group (Experimental): Participant will receive a two-week supply of oral suzetrigine upon discharge. Participant will also receive a 10-pill supply of Oxycodone as a rescue medication.
  Interventions: Drug: oral suzetrigine
- Group B: Oxycodone group (Active Comparator): Participant will receive a two-week supply of oral Oxycodone upon discharge
  Interventions: Drug: oral Oxycodone

INTERVENTIONS:
Drug: oral suzetrigine — patient receives a two-week supply of oral suzetrigine upon discharge
  Arms: Group A: suzetrigine group
Drug: oral Oxycodone — Patient will receive a two-week supply of oral Oxycodone upon discharge
  Arms: Group B: Oxycodone group

SUMMARY:
The purpose this study is determine whether postoperative oral dosage of suzetrigine is effective at controlling postoperative pain and reducing analgesic requirements following primary total knee arthroplasty (TKA) versus a control group of TKA patients receiving postoperative Oxycodone.

DETAILED DESCRIPTION:
The purpose of this prospective, randomized study is to compare the outcomes of two cohorts of patients undergoing primary total knee arthroplasty (TKA) and to determine whether postoperative administration of oral dosage of suzetrigine is effective at reducing postoperative pain versus a control group of patients receiving oral dosage of oxycodone only following primary total knee arthroplasty.

The primary objective will be to compare the amount of postoperative narcotics utilized and postoperative VAS pain levels. The secondary objective will be to compare variables of patient functionality and other patient-reported outcome measures.

The main questions it aims to answer are:

1. What is the efficacy of oral suzetrigine in reducing opioid consumption and postoperative pain following primary total knee arthroplasty?
2. Will the study results demonstrate the effectiveness and safety of oral suzetrigine after primary total knee arthroplasty in reducing postoperative opioid usage while maintaining a similar or better level of pain control when compared to a standard pain control regimen? Researchers will compare suzetrigine to a standard postoperative pain control regimen (Oxycodone) to see if suzetrigine is equivalent or more effective at reducing opioid consumption and postoperative pain following primary total knee arthroplasty.

Participants will:

* be randomized into one of two groups
* undergo a primary TKA
* complete a tracking sheet documenting daily pain medicine usage and VAS pain level for the first 14 days following the TKA
* return to office at 2 weeks and 6 weeks postop for follow-up
* complete additional questionnaires at 2 weeks and 6 weeks postop

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is 21-89 at time of surgery
2. Patient is scheduled to undergo a unilateral primary TKA, secondary to osteoarthritis
3. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization document
4. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 21
2. Patient's primary diagnosis is not osteoarthritis
3. Patient is unable to read and speak English
4. Contraindication or Hypersensitivity to suzetrigine
5. Pregnant or nursing females
6. Patient has taken opioids within the 90 days prior to enrollment

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Daily Opioid Use POD 1-14 | 2 weeks
  Daily opioid use as measured in MME recorded daily for the first two weeks following TKA
total opioid usage over two weeks | 2 weeks
  total daily opioid usage (as measured in MME) for the first 14 days following TKA
Use of supplemental opioid POD 1-14 | 2 weeks
  Average time from initial preop pain control dose to first postop supplemental opioid dose (for participants randomized to Group A, if applicable)
VAS pain score over two weeks | 2 weeks
  VAS (Visual Analogue Scale) pain score measuring highest level of knee pain experienced each day for the first 14 days following TKA. Scale 0-10
Opioid Usage at 6 weeks postop | 6 weeks
  Usage of opioids at 6 weeks postoperatively (Y/N) and if yes, what is daily usage

SECONDARY OUTCOMES:
VAS Pain Score at 6 weeks | 6 weeks
  VAS (Visual Analogue Scale) pain score measuring highest level of knee pain at 6 weeks following TKA. Scale 0-10
KOOS, JR. | preoperatively and 6 weeks (± 2 weeks) postoperatively
  The Knee Injury and Osteoarthritis Outcome Score, Joint Replacement (KOOS, JR) is a survey measuring overall knee health for individuals post total knee arthroplasty (TKA) by evaluating stiffness, pain, function, and activities of daily living. Scoring scale 0-100.
ROM | preoperatively, 2 weeks and 6 weeks (± 2 weeks) postoperatively
  active range-of-motion (ROM) as measured in degrees of extension and degrees of flexion

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Zamora, MD, Study Chair — University of Louisville

IPD SHARING:
Plan to Share IPD: No
Will not share IPD if it is not a requirement

REFERENCES:
- [Result] Mach M, Giba A, Miedziaszczyk M, Bryla A, Szkutnik-Fiedler D. Suzetrigine as a Novel Non-opioid Analgesic Drug in Pain Management: A Review of Clinical Evidence and Therapeutic Perspectives. Cureus. 2025 Aug 22;17(8):e90755. doi: 10.7759/cureus.90755. eCollection 2025 Aug. PMID 40862032
- [Result] The Lancet Regional Health-Americas. Opioid crisis: addiction, overprescription, and insufficient primary prevention. Lancet Reg Health Am. 2023 Jul 12;23:100557. doi: 10.1016/j.lana.2023.100557. eCollection 2023 Jul. No abstract available. PMID 37497399
- [Result] Robert M, Jouanjus E, Khouri C, Fouilhe Sam-Lai N, Revol B. The opioid epidemic: A worldwide exploratory study using the WHO pharmacovigilance database. Addiction. 2023 Apr;118(4):771-775. doi: 10.1111/add.16081. Epub 2022 Nov 22. PMID 36331523